CLINICAL TRIAL: NCT02822131
Title: The Effect of Dietary Phosphate Intake on Blood Pressure Regulation and Renal Sodium Chloride Excretion in Healthy Male Volunteers
Brief Title: Phosphate in Blood Pressure Regulation
Acronym: Phos-RR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Nilufar Mohebbi, PD Dr. med., University of Zurich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: Phos-RR
Record Dates: First submitted 2016-04-08; First posted 2016-07-04 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — sodium phosphate; Sevelamer; Sodium Bicarbonate; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low phosphate (Other): low phosphate will be induced by low phosphate diet and additional treatment with oral phosphate binder sevelamer.
  Interventions: Drug: sevelamer, sodium bicarbonate, sodium chloride
- high phosphate (Other): high phosphate diet will be induced by oral supplementation with sodium phosphate.
  Interventions: Dietary Supplement: sodium phosphate

INTERVENTIONS:
Dietary Supplement: sodium phosphate
  Arms: high phosphate
Drug: sevelamer, sodium bicarbonate, sodium chloride
  Arms: low phosphate

SUMMARY:
High dietary phosphate intake in the general population is associated with a higher risk for developing kidney disease and cardiovascular disease with an increased overall mortality. Whereas the effects of high phosphate intake on general health become clearer, almost nothing is known about underlying mechanisms. More recently, the investigators and others found in animal models that FGF23 stimulates the renal NaCl cotransporter NCC, the target of thiazide diuretics, and that increased NCC activity may increase blood pressure. The investigators could also show that increasing dietary phosphate intake in mice, increases FGF23 and NCC activity within 3 days. Thus, the objective of this single-centre observational cross-over study including 20-45 year old healthy male probands is to elucidate the role of dietary phosphate on blood pressure regulation and renal handling of sodium chloride in healthy subjects. Further the impact of dietary phosphate intake on the regulation of phosphaturic hormones and other factors regulation blood pressure will be investigated. In addition, the investigators will examine whether phosphate intake modulates gut microbiome composition. The primary outcome in this study is the change in blood pressure in healthy subjects on low-phosphate diet compared to healthy subjects on high-phosphate diet. In addition, to assess changes in NCC activity as the main mechanism of phosphate-sensitive blood pressure regulation, renal sodium chloride excretion after administration of hydrochlorothiazide will be measured. The secondary outcomes of this study are: changes in renal phosphate, calcium and potassium excretion, changes in phosphate regulation hormones such as 25-OH-Vit. D, 1,25-(OH)2-Vit. D, PTH, FGF23, dopamine in plasma and urine, changes in plasma and urinary aldosterone levels, changes in sodium/chloride-cotransporter NCC and NaPi-IIa assessed from urinary exosomes, and changes in stool phosphate excretion and gut microbiome composition.

ELIGIBILITY:
Inclusion Criteria:

* 20-45 year old healthy male subjects

Exclusion Criteria:

* - Kidney disease (defined by eGFR < 90 ml/min or microalbuminuria (> 30mg/d))
* Diabetes mellitus
* Hypertension (RR > 140/85 mmHg)
* Hypotension (RR < 90/60 mmHg)
* any regular medication
* non-Western type diet e.g. vegetarian, vegan etc.
* History of kidney stones
* Allergy to sulphonamides or penicillins
* Hereditary fructose intolerance
* known hypersensitivity or allergy to class of drugs used in this study
* Glaucoma
* Vitamin D deficiency (< 20 ng/ml)
* Hyper- or Hypoparathyroidism
* Hypo- or hyperaldosteronism
* Participation in any other study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | 5 days
Change in renal sodium chloride excretion | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Nephrology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No